CLINICAL TRIAL: NCT01271491
Title: The Genetics of Respiratory Failure in Bronchiolitis
Status: Completed | Type: Observational
Sponsor: Connecticut Children's Medical Center (Other)
Collaborators: UConn Health (Other)
Responsible Party: Principal Investigator, Christopher Carroll, MD, Associate Professor of Pediatrics, Connecticut Children's Medical Center
Other Study IDs: 10-097
Record Dates: First submitted 2010-11-09; First posted 2011-01-06 (Estimated); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Bronchiolitis
Keywords: Pediatric
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva and blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Children hospitalized in the ICU with bronchiolitis
- Controls: Children hospitalized in the general ward with bronchiolitis

SUMMARY:
Bronchiolitis is a potentially severe infection of the airway in infants and children, and among the most frequent diagnoses leading to pediatric intensive care unit admission in infants. This acute infection is caused by an array of viruses, but respiratory syncytial virus (RSV) is the most frequently implicated. The majority of infants hospitalized with bronchiolitis are previously healthy, and half of infants intubated and mechanically ventilated for respiratory failure due to RSV bronchiolitis have no previously identified risk factors. It is likely, therefore, that other factors, particularly genetic heterogeneity of the host, contribute to disease severity. However, no previous study has investigated the association of genetic variants with respiratory failure in children with bronchiolitis. Several categories of candidate genes have emerged as potentially important in the pathogenesis of the disease. Specifically, genetic polymorphisms of surfactants, pattern recognition receptors, receptor adhesion molecules, and cytokines have been examined. The aim is to evaluate these polymorphisms to determine their association with respiratory failure in a cohort of more severely ill children with bronchiolitis.

DETAILED DESCRIPTION:
We propose to conduct a prospective observational study of infants and children admitted with bronchiolitis to determine if genetic polymorphisms in a number of likely candidate immune response related genes are positively associated with respiratory failure in this population. Respiratory failure will be defined as requiring intubation and mechanical ventilation. We plan to enroll two groups of children, those admitted to the ICU with respiratory failure due to bronchiolitis (cases) and those children admitted to the ward with less severe bronchiolitis infection (controls). In special circumstances, we will also enroll pairs of twins who are hospitalized with bronchiolitis (in the ICU or the ward), for whom either one or both twins do not meet inclusion criteria as a case or a control and/or for whom we are not able to obtain a DNA blood sample while hospitalized (twin inpatient population).

Demographic data, and data regarding the hospital treatments and course of these children will be collected. Blood, saliva or sputum for genotyping will also be obtained. If a patient enrolled as a control needs to be intubated, these children cannot be control patients, but instead would be considered cases.

We propose to compare a population of 100 children with respiratory failure due to bronchiolitis to a population of 100 children with bronchiolitis without respiratory failure. Clinical characteristics and genetic markers will be compared. We will also compare clinical characteristics and genetic markers of any twin pairs who are enrolled.

ELIGIBILITY:
Inclusion Criteria, cases:

* admission to the ICU with a primary diagnosis of bronchiolitis
* endotracheally intubated and mechanically ventilated with respiratory failure due to bronchiolitis
* age less than 2 years

Exclusion Criteria, cases:

* pre-existing chronic disease including:

  1. bronchopulmonary dysplasia
  2. congenital heart disease
  3. immune deficiency
* requiring an additional venopuncture for blood collection for genotyping

Inclusion Criteria, controls:

* admission to the hospital with a primary diagnosis of bronchiolitis
* age less than 2 years

Exclusion Criteria, controls:

* pre-existing chronic disease including:

  1. bronchopulmonary dysplasia
  2. congenital heart disease
  3. immune deficiency
* requiring an additional venopuncture for blood collection for genotyping
* requiring non-invasive positive pressure ventilation or high flow nasal cannula
* requiring intubation and mechanical ventilation during the hospitalization

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children hospitalized with bronchiolitis
Sampling Method: Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2010-11; Primary Completion 2018-04 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Respiratory Failure | 2 years
  The primary end point is respiratory failure.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher L Carroll, MD, MS, Principal Investigator — Connecticut Children's Medical Center
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No